CLINICAL TRIAL: NCT00090376
Title: Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 3 Arm, 12-Month Study to Evaluate the Effects of GPI 1485 on Erectile Function in Patients Undergoing Bilateral Nerve-Sparing Radical Retropubic Prostatectomy for Prostatic Carcinoma
Brief Title: Evaluate the Effects of GPI 1485 on Erectile Function Following Bilateral Nerve-Sparing Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Symphony Neuro Development Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0501-0202
Record Dates: First submitted 2004-08-25; First posted 2004-08-30 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Impotence; Prostate Cancer
Keywords: Erectile Dysfunction; Impotence; Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — GPI 1485

INTERVENTIONS:
Drug: GPI 1485

SUMMARY:
In this phase II study, an investigative (not approved by the FDA) drug called GPI 1485 is being assessed to see if it can help preserve erectile function after prostatectomy.

DETAILED DESCRIPTION:
This drug has been tested in animals, and was shown to protect nerves from damage and to regrow damaged nerves in these animal studies. Participants will receive either GPI 1485 or a placebo (inactive pill). Participants will begin study medication 3 full days prior to their scheduled surgery.

GPI 1485 will be supplied as an oral tablet formulation to men who are candidates for bilateral nerve-sparing prostatectomies. Participants randomly assigned to receive GPI 1485 will be required to take four tablets four times a day by mouth.

GPI 1485 matching placebo will also be supplied as an oral tablet formulation. Participants randomly assigned to placebo will be required to take 4 placebo tablets four times a day by mouth.

Viagra® will be supplied as oral tablets beginning 1 month post-surgery. Patients can begin Viagra® 1 month post-surgery and may continue use until the end of the study, as needed.

The duration of this study is 12 months which includes 5 office visits to your doctor in addition to the surgery day. During this study you will also have other clinical evaluations including a physical exam, blood work, ECG (tracing of your heart rhythm) and urinalysis.

Participants enrolled in this study will also carry a handheld diary that is loaded with special protocol-specific software, which will be referred to as the patient experience diary (PED). Over the duration of this study, participants will complete their questionnaires and answer questions about their medication compliance in the electronic PED.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of localized prostate carcinoma and scheduled to undergo curative surgical resection via bilateral nerve sparing procedure.
2. Localized prostate cancer is defined as:

   * Gleason score <=7 (<=3 + <=4)
   * PSA <=10 off of finasteride (Proscar®) and dutasteride (Avodart®)
   * <=T2a stage disease
3. Motivated males, 40 to 69 years of age inclusive, and in the opinion of the investigator, are currently in a monogamous, sexually active relationship.
4. Males that have erectile function (EF) (without the use of pharmacotherapy within 30 days prior to screening assessment).
5. EF is defined as a score of >=26 on the EF domain of the IIEF questionnaire based on patient experiences over the 4 weeks prior to biopsy.
6. Body Mass Index (BMI) within the 18-34.9 kg/m2 range.
7. Able to swallow whole tablets equivalent to capsule size 0.
8. Available for protocol-specified visits and procedures.
9. Informed written consent must be provided prior to any study-specific procedures.

Exclusion Criteria:

1. Recent history, within 6 months before screening, of drug or alcohol abuse.
2. History of peripheral neuropathy.
3. History of acute or chronic depression that in the opinion of the investigator may interfere with protocol-specified efficacy measurements.
4. History of diabetes that requires use of insulin or oral hypoglycemic agents, myocardial infarction, or cerebrovascular accident.
5. History of spinal trauma or surgery to the brain or spinal cord.
6. Any medical disability or laboratory abnormality (e.g., serum creatinine > 2.0 mg/dL) that, in the opinion of the Investigator, may interfere with the protocol-specified safety and efficacy measurements, present an unacceptable risk to the patient's well-being, or compromise the patient's ability to provide informed consent.
7. History of pelvic radiation therapy (external beam radiation or brachytherapy).
8. Concomitant use of hormonal therapy, vasodilators (nitrates), dutasteride (Avodart®) or finasteride (Proscar®) within the 30 days prior to biopsy and throughout the study.
9. Concomitant use of therapeutic agents to treat ED other than those specified in the protocol is not permitted starting at least 30 days prior to biopsy and continuing throughout the study.
10. Previous exposure to GPI 1485 (previously AMG-474-00).
11. Treatment with an investigational agent within the 30 days before screening or scheduled to receive an investigational agent other than that specified by this protocol during the course of this study.
12. Any contraindication to Viagra® use
13. Unable to stop the use of inducers or inhibitors of cytochrome P450 (CYP) 3A4 from Baseline until the end of the study.

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Favit-Van Pelt, MD, PhD, Study Director — Eisai Inc.
Locations (25):
- United States (25):
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Center for Urological Research, La Mesa, California
  - Stanford University Medical Center, Stanford, California
  - Connecticut Surgical Group, Hartford, Connecticut
  - Connecticut Urological Research at Grove Hill, New Britain, Connecticut
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Vattikuti Institute for Urology, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - PPS Clinical Research, St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Urology Associates, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Carolinas Health Care System McKay Urology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Urological Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington